CLINICAL TRIAL: NCT02371993
Title: Asthma in the Elderly: A Study of Choline Supplementation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C. (Other)
Responsible Party: Principal Investigator, Michele Columbo, M.D., Principal Investigator, Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F/N-R15-3427B
Record Dates: First submitted 2015-02-10; First posted 2015-02-26 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Asthma in the Elderly
MeSH Terms: interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Choline 650 mg twice daily (Experimental): See above
  Interventions: Dietary Supplement: Choline; Other: Placebo
- Placebo (Placebo Comparator): See above
  Interventions: Dietary Supplement: Choline; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Choline
Other: Placebo

SUMMARY:
Asthma in the elderly is poorly understood, as most studies have not included this patient group. In a previous study of adults with asthma, choline supplementation had a positive effect on asthma symptoms and allowed to decrease asthma pharmacologic treatment. The present study is a randomized, double-blind, placebo-controlled, cross-over study of choline supplementation. The investigators will study the effect of choline 650 mg taken orally twice daily x 6 weeks versus placebo on asthma symptom scores (Asthma Control Test) and spirometric values (FEV1, FEV1/FVC, FEF25-75%). The investigators will also look at the effect of choline supplementation on peripheral blood eosinophils, serum immunoglobulin E (IgE) and homocysteine levels.

ELIGIBILITY:
Inclusion Criteria:

* Asthma

Exclusion Criteria:

* No history of smoking more than 10 pack/years,
* no gastrointestinal cancers,
* no liver or kidney disease,
* no bipolar disorder.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Effect of choline supplementation on asthma symptoms measured by the Asthma Control Test | six weeks
Effect of choline supplementation on spirometric values (FEV1, FEV1/FVC, FEF25-75%) | six weeks

SECONDARY OUTCOMES:
Effect of choline supplementation on peripheral blood eosinophils | six weeks
Effect of choline supplementation on serum IgE | six weeks
Effect of choline supplementation on serum homocysteine levels | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michele Columbo, M.D., Principal Investigator — Rohr and Columbo Asthma, Allergy and Immunology Specialists
Locations (1):
- Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C., Bryn Mawr, Pennsylvania, United States

REFERENCES:
- [Derived] Columbo M, Rohr AS. Asthma in the elderly: the effect of choline supplementation. Allergy Asthma Clin Immunol. 2016 Mar 11;12:15. doi: 10.1186/s13223-016-0121-5. eCollection 2016. PMID 26973701